CLINICAL TRIAL: NCT03149159
Title: An Investigator-Initiated Trial of Combined Ipilimumab, Nivolumab and Stereotactic Radiation in Patients With Metastatic Clear-Cell RCC (ccRCC) Who Have Failed Treatment With Single-Agent Nivolumab
Brief Title: Investigator-Initiated Trial of Combined Ipilimumab, Nivolumab and Stereotactic Radiation in Patients With Metastatic Clear-Cell RCC (ccRCC) Who Have Failed Treatment With Single-Agent Nivolumab
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study is withdrawn due to feasibility issues.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102576; CA209-927 (Other Grant/Funding Number: BMS)
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Clear Cell Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab + Ipilimumab + SRT (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Radiation: Steriotactic radiation therapy

INTERVENTIONS:
Drug: Nivolumab — Nivolumab will be given every 21 days for the first 12 weeks at a dose of 3mg/kg. After 12 weeks, the dose will be 240mg and will be given every 14 days.
  Other Names: opdivo
Drug: Ipilimumab — Ipilimumab will be given at a dose of 1mg/kg every 21 days for up to 12 weeks.
Radiation: Steriotactic radiation therapy — The dose of radiation will be 6 Gy daily x 5 days. Radiation will be given between the first and second doses of ipilimumab plus nivolumab.

SUMMARY:
The purpose of this study is to see if continued nivolumab with the addition of ipilimumab plus hypo-fractionated stereotactic radiation (sTR) of a single lesions results in partial or complete responses in patients with metastatic ccRCC who fail initial treatment with single agent nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic ccRCC.
* Age 18 years and older
* ECOG 0-1
* Progressive disease after treatment with single-agent nivolumab
* Life expectancy at least 3 months
* Presence of measurable disease per RECIST 1.1 criteria
* Presence of a metastatic lesion greater than 1 cm in size that is amenable to radiation treatment
* Adequate organ system function
* WOCBP and men who are sexually active with WOCBP must agree to use appropriate method(s) of contraception.

Exclusion Criteria:

* Patients are excluded if they have active brain metastases or leptomeningeal metastases (exceptions outlined in the protocol).
* Active, known or suspected autoimmune disease, such as systemic lupus erythematosus, that require treatment with immune suppressing drugs.

Note: Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger

* Presence of a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalents) or other immunosuppressive medications within 14 days of study drug administration.

Note: Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

* Unstable angina or uncontrolled congestive heart failure
* Uncontrolled hypercalcemia
* Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Presence of other malignant diseases, except non-melanoma skin care
* History of allergy to study drug components.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Anti-cancer treatment including surgery, radiotherapy, chemotherapy, other immunotherapy, or investigational therapy within 14 days of registration.
* Women must not be pregnant or breastfeeding. WOCBP must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to registration.
* Any other medical condition for which treatment with ipilimumab or nivolumab would be medically contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with a partial or complete response | 12 weeks
  The response rate of combined ipilimumab and nivolumab plus STR will be determined using irRECIST criteria.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  PFS will be determined from the onset of treatment to the time of documented disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lilly, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No